CLINICAL TRIAL: NCT01435291
Title: Prospective Pharmacokinetic and Pharmacogenetic Analysis of Advagraf After Transplantation
Brief Title: AADAPT - Analysis of Advagraf Dose Adaptation Post Transplantation
Acronym: AADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-PP-07
Record Dates: First submitted 2011-09-15; First posted 2011-09-16 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-08

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf (Experimental)
  Interventions: Drug: Advagraf Capsule
- Prograf (Active Comparator)
  Interventions: Drug: Prograf Capsule

INTERVENTIONS:
Drug: Advagraf Capsule — Other Names:
  * FK506E
  * MR4
  * tacrolimus modified/prolonged release Drug: MPA Solution for infusion and per os Other Name: Mycophenolate Mofetil or Mycophenolic Acid Drug: Basiliximab IV infusion Other Name: Simulect Drug: Corticosteroids per os Other Name: Methylprednisolone or equivalent
  Arms: Advagraf
Drug: Prograf Capsule — Other Names:
  * FK506E
  * MR4
  * tacrolimus Drug: MPA Solution for infusion and per os Other Name: Mycophenolate Mofetil or Mycophenolic Acid Drug: Basiliximab IV infusion Other Name: Simulect Drug: Corticosteroids per os Other Name: Methylprednisolone or equivalent
  Arms: Prograf

SUMMARY:
A pharmacokinetics and pharmacogenetics study to complement the current knowledge of tacrolimus prolonged release (Advagraf®) in the immediate post-transplantation period and at steady-state (M3 post transplantation) and to improve the optimal dose of Advagraf® based on tacrolimus AUC estimated by two Limited Samples Strategies during the first 3 months after renal transplantation.

Data obtained with tacrolimus prolonged release will be compared with those of tacrolimus immediate release (Prograf®)

DETAILED DESCRIPTION:
Multicentre open-labeled randomized pharmacokinetic (PK) and pharmacogenetic (PG) study to compare Advagraf and Prograf immediate post-transplantation (Day 8) and steady-state (Day 84) systemic exposure.

Tacrolimus PK profile, tacrolimus systemic exposure assessed by Limited Samples Strategies (LSS) (i.e.: Bayesian estimators (BE) and Multilinear Regressions (MLR)), and impact of CYP3A5 and ABCB1 genetic polymorphisms on tacrolimus PK will also be determined to improve the optimal dose of Advagraf® for kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients aged between 18 to 70
* Primary renal transplantation
* Cadaver or living transplantation or living (non HLA identical) donor with compatible ABO blood type.
* absence of anti-LHA antibodies in lymphocytotoxicity and Luminex
* Negative cross-match in cytotoxicity
* Negative pregnancy test for female patients of childbearing potential, and agreement to practice effective birth control during the study

Exclusion Criteria:

* Combined transplantation
* Renal bigraft
* History of any other transplantation
* Receiving a graft from a non-heart-beating donor.
* Requiring ongoing dosing with a systemic immunosuppressive drug prior to transplantation
* Patient who received within one month prior to study an inductor of CYP50 3A or requiring during the study an inhibitor of CYP50 3A or of P-gp.
* Significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer
* Subject or donor known to be HIV positive
* Active viral hepatitis (VHB, VHC) at randomisation
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, corticosteroids, or mycophenolate mofetil or any of the product excipients
* Diagnosis of new-onset malignancy prior to transplantation, with the exception of basocellular or squamous cell carcinoma of the skin which had been treated successfully.
* Current participation in any other clinical study
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the study
* Patient not able to comply with the study procedures
* Breast-feeding mother

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
AUC 0-24h of tacrolimus at Day 8 and Day 84 | 3 months

SECONDARY OUTCOMES:
AUC 24h of tacrolimus using limited samples strategies (LSS) at Day 8 and Day 84 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth CASSUTO, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (4):
- France (4):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Nice, Nice
  - CHU de Rangueil, Toulouse
  - CHRU Tours Hôpital Bretonneau, Tours